CLINICAL TRIAL: NCT02043795
Title: Drug Impregnated Bioabsorbable Stent in Asian Population Extremity Arterial Revascularization (DISAPEAR Study)
Acronym: DISAPEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013/539/C
Record Dates: First submitted 2013-10-29; First posted 2014-01-23 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Critical Limb Ischemia
Keywords: Bioresorbable Vascular Scaffold System; Percutaneous Transluminal Angioplasty; Stent
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated with BVS (Other): Symptomatic patients would be screened with a duplex ultrasound as per clinical practice prior to intervention. After informed consent for a standard angiography/intervention, the patient will undergo a planned intervention under general or local anaesthesia in an angiographic facility.
  Interventions: Device: BVS, Abbott Vascular

INTERVENTIONS:
Device: BVS, Abbott Vascular — The aim of this study is to study the safety and clinical efficacy of a novel Bioabsorbable Everolimus Eluting Bioresorbable Vascular Scaffold System (BVS, Abbott Vascular).
  Other Names: Bioresorbable Vascular Scaffold System

SUMMARY:
The aim of this study is to study the safety and clinical efficacy of a novel Bioabsorbable Everolimus Eluting Bioresorbable Vascular Scaffold System (BVS, Abbott Vascular) in subjects with critical limb ischemia (CLI) following percutaneous transluminal angioplasty (PTA) of the tibial arteries.

DETAILED DESCRIPTION:
Background

Currently, DM foot admissions account for up to 2% of all admissions in CGH, with up to 50% of patients with peripheral vascular disease (PVD). CGH Vascular service performs 100-150 peripheral angioplasties for limb ischaemia per 6 months, the majority of which are for limb salvage procedures. The angioplasty procedure is performed below the knee (BTK) and the BTK vessels are involved in more than 80% of the time. Restenosis is common in peripheral interventions.

In the recently published DESTINY trial, the superiority of Everolimus DES (XIENCE, Abbott Vascular) was proven over BMS (Bare Metal Stents). This landmark study suggests that for short lesions in the BTK segment, DES improved patency rates and reduced the need for re-interventions for restenosis.

Re-interventions for previously stented arteries are technically difficult. In the coronary bed, the Bioabsorbable stents have been developed to provide the functions of a drug eluting stent but yet provide a temporary scaffold to allow the vessel to heal. The absence of a permanent metallic implant in the vascular tissue may facilitate any required re-interventions on the target vessel / lesion or side branches either by percutaneous or surgical means, thus enabling a broader range of treatment options after bioresorption of the scaffold. In addition, unlike permanent metal implants, polymeric implants do not cause imaging artifacts during non-invasive CT or MR evaluation providing additional benefit

Rationate and justification for the study

The safety of the BVS has already been demonstrated in man in the Coronary Bed. It is currently CE marked for this indication.

In the ABSORB Cohort A Study, it showed excellent long term clinical outcomes with low MACE rates out to 4 years with absence of any target lesion revascularization, Q-wave myocardial infarction, and scaffold thrombosis. Cohort B confirms these findings out to 1 year; including patency comparable to XIENCE V. Absorb BVS thus performs all the functions of a drug-eluting stent while offering future potential benefits resulting from the absence of a permanent metallic implant.

An optimal post procedural follow-up imaging technique is as yet uncertain for this stent. Assessment of conventional stents with CT angiography has been limited by streak and susceptibility artefact on MRA. Doppler Ultrasound is known to be time intensive. Hence, if MRA or CTA proof to be accurate modalities for evaluation, it would be easier for follow-up and evaluation of these patients.

The aims of this study are:

1. to study which non-invasive imaging modality would be most appropriate in follow-up for Bioabsorbable Everolimus Eluting Bioresorbable Vascular Scaffold System (BVS, Abbott Vascular) patency deployed in subjects with critical limb ischemia (CLI) following percutaneous transluminal angioplasty (PTA) of the tibial arteries. The aim is to establish stent patency as well as imaging features of the stent.
2. to investigate the effects of percutaneous transluminal angioplasty using Bioabsorbable Vascular Scaffold (BVS) in patients with Critical Limb Ischaemia CLI) and Below the Knee (BTK) lesions in an Asian Population. One of the side arms of the study is to establish imaging features of this new stent system with Doppler ultrasound, CT angiography and MR angiography. The study aims to establish stent patency, as well as imaging features of stent as it bio reabsorbs.

Study design

The study will prospectively collect consecutive cases treated with BVS for patients with CLI and BTK lesions recruited over a 2 year period and followed up for 1 year. The results of these patients will be compared to a similar historical cohort consecutively treated with XIENCE DES (metallic Drug Eluting Stents, Abbott Vascular).

This pilot study will involve recruitment of 12 patients x 1 year followed by another year of post implantation follow-up. If feasible, the recruitment will be extended to another year for another 12 patients giving a total of 24 patients.

Patients not on chronic antiplatelets therapy should receive a loading dose of Plavix 300 mg and Aspirin 300 mg started 6 to 72 hours prior and not later than 1 hour after the procedure. Pre procedure clinical assessment including pulses and Transcutaneous O2 measurement around the affected wound. In the absence of a wound, this will be performed on the dorsum of the foot. Demographic data including comorbidities, medication history, Rutherford class will be recorded.

Symptomatic patients would be screened with a duplex ultrasound prior to intervention. After informed consent for a standard angiography/intervention, the patient will undergo a planned intervention under general or local anaesthesia in an angiographic facility. Either antegrade or retrograde approach is allowed. After common femoral artery sheath access, a diagnostic angiogram will be performed as per any standard angioplasty procedure. 2 plane angiography of the target lesions will be performed. Of note will be the lesion characteristics like length, location, and degree of stenosis and calcification. Degree of runoff will also be assessed on angiography. If the 2 plane angiography confirms > 50% stenosis or occlusion, the patient will be eligible for BVS. The target vessel chosen should preferably be but should not limited to, the wound relate artery in accordance to the angiosome concept. There should at least be one vessel runoff to the foot.

After angiographic assessment for suitability for BVS, heparin 2500 to 5000 IU will be administered intra-arterially as per standard angioplasty according to body weight. The stenosis of occlusion will be crossed (true lumen or subintimal crossing is allowed) with a guidewire of choice and pre-dilatation with a balloon catheter will be performed. Pre-dilatation should be in accordance with manufacturer guidelines an should not extend beyond the proposed treated segment

Post intervention angiography will subsequently be performed to assess the success of treatment repeat balloon inflation is allowed. Any residual stenosis and the degree of stenosis at the end of the intervention will also be recorded. Post dilatation should be confined to the previously scaffolded area and not exceed manufacturer recommendations with respect to size. Subsequent treatment of the runoff tibial vessels is allowed.

Post procedure, standard post angioplasty regimes will be followed. Patients will be started on supplementary Clopidogrel (Plavix) 75 mg once a day together with Aspirin 100mg once a day i.e. dual antiplatelets for 6month post intervention followed by Aspirin for life unless contraindicated.

Clinical follow-up will be performed immediately post procedure at 1 month, 6 months and 1 year post intervention. Assessment of the pulse, clinical patency will be performed at each visit. TCOMs will be performed at 6 and 12 months. Duplex ultrasound to assess for re-stenosis will be performed at 6 and 12 months, while CT angiography and MR angiography will be performed at 12-month post-procedure.

ELIGIBILITY:
Criteria for Recruitment

At the investigator site, the investigators will recruit patients in accordance to the study protocol, local regulatory requirements, and the ICH-GCP guidelines. When a patient is identified, he/she will be informed about the study. The study will be fully explained to the patient including study objectives, methods, anticipated benefits/risks and discomforts he or she may experience. Summary of this information will be provided in writing using the Informed Consent Form. Patients will be given the opportunity to clarify any issues/questions with the investigator and given adequate time to consider participating in the study or not. Signed and dated informed consent of the patients will be obtained before the commencement of any study related procedures.

Inclusion Criteria:

* Stenotic (> 50%) or occlusive atherosclerotic disease of the infrapopliteal arteries
* A maximum of 2 target lesions in one or more infrapopliteal vessels
* Minimum of 1mm overlap of stents
* Reference vessel diameter should be 2-4.0 mm
* Symptomatic critical limb ischemia (Rutherford 4, 5, 6)
* The patient must be > 21 years of age
* Life-expectancy of more than 12 months
* The patient has no child bearing potential or negative serum pregnancy test within 7 days of the index procedure
* The patient must be willing and able to return to the appropriate follow-up times for the duration of the study
* The patient must provide written patient informed consent

Exclusion Criteria:

* Patient refusing treatment
* The reference segment diameter is not suitable for available stent design
* Unsuccessfully treated (>50% residual stenosis) proximal inflow limiting arterial stenosis
* Untreatable lesion located at the distal outflow arteries
* Lesion location requiring kissing stent procedure
* The patient has a known allergy to heparin, Aspirin or other anticoagulant/anti-platelet therapies or a bleeding diatheses or is unable, or unwilling, to tolerate such therapies.
* The patient takes Phenprocoumon (Marcumar).
* The patient is currently breast-feeding, pregnant or intends to become pregnant.
* Subject is receiving immunosuppression therapy, or has known serious immunosuppressive disease (e.g., human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., systemic lupus erythematosus, etc.) The patient should also not receive inhibitors of CYP3A (such as Itraconazole, and Erythromycin), or inducers of CYP3A (such as Rifampin) within 90 days following the procedure.
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure to the target vessel

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in Re-stenosis rates between 6 months and 12 months | 6 months and 12 months
  defined at stenosis >=50% of the treated segment on duplex ultrasound, CT angiography or MR angiography

SECONDARY OUTCOMES:
Change in Mean Transcutaneous oxygen measurement (TCOMs) between 6 months and 12 months | 6 and 12 months
  Change in Mean Transcutaneous oxygen measurement (TCOMs)
Change in Amputation free survival between 6 months and 12 months | 6 months and 12 months
Change in Freedom from Target lesion revascularization between 6 months and 12 months | 6 and 12 months
Change from baseline in Rutherford class at 6 months and 12 months | Baseline, 6 and 12 months
Number of Participants with major adverse limb events (MALE) | within 1 year
  Freedom from major adverse limb events (MALE) within 1 year
Number of Participants with Peri-procedural death (POD) | within 30-day
  Freedom from peri-procedural (30-day) death (POD)

OTHER OUTCOMES:
Sensitivity and specificity of each imaging modality | 1 year
  Imaging features of the Bioabsorbable Everolimus Eluting Bioresorbable Vascular Scaffold System would be evaluated on the various imaging modalities, like possible streak artefacts on CT scan and susceptibility on MR. Sensitivity and specificity of each imaging modality will be compared with one another as well as those in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kum, MD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore